CLINICAL TRIAL: NCT02826460
Title: Psychosocial Predictors of Posttransplant Adherence and Outcomes
Brief Title: Psychosocial Risks in Liver Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 14-1874
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: End Stage Liver Disease
Keywords: Transplant; Adherence
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver Transplant Recipients

SUMMARY:
A retrospective chart review in which the information in the standard psychosocial evaluations done pre-transplant for liver transplant recipients will be coded, recorded, and correlated with posttransplant outcomes of the same recipients. Evaluated outcomes include rejection episodes and adherence to tacrolimus, calculated through the MLVI (Medication Level Variability Index). The researchers will evaluate the degree to which both single elements in the evaluation as well as a cumulative score derived by a structured review of the chart using the Stanford Integrated Psychosocial Assessment for Transplantation (SIPAT) model can predict posttransplant outcomes.

DETAILED DESCRIPTION:
The research team will perform a chart review and extract data without identifiers from paper charts and electronic charts and data tracking system. This data will be obtained from OTTR /EPIC as well as paper charts if needed. Those charts will be accessed to obtain demographic data (age, gender, income, employment status, marital/relationship status, insurance payer); transplant specific data (primary diagnosis, transplant year, tacrolimus blood levels, rejection episodes (yes/ no and number of), graft loss (yes/no), re-transplantation (yes/no); related medical data (creatinine levels, dialysis dependence (yes/no), ICD diagnoses; and psychosocial variables (social worker risk assessment before transplant, presence of social and family support, conviction history (yes/no), psychiatric history (diagnoses yes/no).

Variables will be obtained from the psychosocial pretransplant evaluation write-up (which in different years was attached to OTTR or EPIC datasets, or may be present in paper form, and from electronic datasets (OTTR / EPIC).

The data extraction as well as dataset building and data entry will be performed in office spaces at ISMMS. No patient contact is anticipated for this study. The predictive model will include evaluations of single variables as well as an evaluation of the predictive ability of a pre-defined scoring system (the SIPAT) which will be applied to existing data.

ELIGIBILITY:
Inclusion Criteria:

* Received a liver transplant in the year 2012 or earlier
* Received Tacrolimus
* Had at least 3 Tacrolimus blood tests
* Received their transplant at RMTI

Exclusion Criteria:

* Patients who received more than 1 solid organ transplant
* Patients who were not prescribed Tacrolimus
* Patients who died within the first year after transplant
* Patients with cognitive impairment

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whose information is available to RMTI, who received a liver transplant in the year 2012 or earlier, who received tacrolimus, and who had at least 3 tacrolimus blood tests, are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Rejection | 2 years
  Number of Rejections confirmed by biopsy

SECONDARY OUTCOMES:
Medication Level Variability Index (MLVI) | 2 years
  MLVI is a measure of medication adherence

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shemesh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinia, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No